CLINICAL TRIAL: NCT05852821
Title: The 5 Repetitions Sit-to-stand Test, Carried Out Remotely Via Videoconference, in Patients With COPD: Is There a Learning Effect?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: e-EVAL
Record Dates: First submitted 2023-04-27; First posted 2023-05-10 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Chronic Respiratory Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- remote 5STS through videoconference (Experimental)
  Interventions: Other: 5STS remote assessment via videoconference

INTERVENTIONS:
Other: 5STS remote assessment via videoconference — Patients will be asked to perform several times the 5STS test, from their home through videoconference, on 3 occasions (day 1, 24h later and 1month later).

SUMMARY:
The purpose of this clinical study is to determine if a learning effect exists when the 5STS is assessed remotely via videoconference in patients with COPD.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR) is an essential therapy for improving exercise tolerance and quality of life in patients with chronic respiratory disease. It is now available remotely thanks to advances in information and communication technologies. Pulmonary telerehabilitation facilitates care access for patients living far from specialized centers. It requires, for a complete and coherent transposition, to be able to evaluate the patients remotely in order to measure the evolution of their functional capacities and to ensure their follow-up. Among the tests already implemented at home and remotely via video-conference, the 5-repetition sit-to-stand test (5STS) is the most suitable. This test requires only a short time to perform, little space and no specific equipment. However, two major limits remain to be checked before being able to consider its remote and routine implementation. First of all, it is important to study its feasibility. Moreover, like other functional tests, it raises the question of a possible learning effect (LE). In the perspective of a current use of the 5STS remotely, it is therefore also essential to assess the existence of a potential LE which would condition the methods of administering the test and its interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Obtaining oral informed consent after a minimum reflection period of 24 hours
* Patient with internet access at home and a tool allowing the realization of a videoconference (smartphone or computer)

Exclusion Criteria:

* Patients who had a recent exacerbation (less than 4 weeks)
* Patients physically unable to get up from a chair and sit down without help
* Patients with significant and unstable cardiovascular disease
* Any acute or chronic pathology (orthopedic, neurological, psychiatric or causing a major cognitive disorder) limiting the performance of a functional test
* Inability or difficulty using digital tools
* Subjects in a period of relative exclusion compared to another protocol
* Adults protected by law or patient under guardianship or curatorship
* Subjects deprived of liberty by a judicial or administrative decision
* Current or planned pregnancy during the study period
* Pregnant or breastfeeding women
* Patients not affiliated to a French social security scheme or not benefiting from such a scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
the variation in time of 5STS between first assay and fifth assay during the first visit (V1). | 1 day

SECONDARY OUTCOMES:
the variation in time of 5STS between each trial at the first visit (V1). | 1 day
the variation in time of 5STS between the first visit (V1) and the second visit (V2). | 2 days
the variation in time of 5STS between the second visit (V2) and the third visit (V3). | 1 month
The reproducibility of the remote test | 1 month
  Reproducibility is objectified by the test-retest reliability between two trials of the same series (first and fifth trials of V1) and between two series (V1-V2; V2-V3; V1 -V3).
The number of tests not carried out | through study completion, an average of 1 year
Patient satisfaction | 1 month
  Satisfaction will be assessed with a questionnaire at the end of visit 3.
The number of connection failures | through study completion, an average of 1 year
The number of patients excluded because of the video-conference tool | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nelly HERAUD, Study Director — Director of research
Locations (1):
- Clinique du Souffle la Vallonie, Lodève, France

IPD SHARING:
Plan to Share IPD: No